CLINICAL TRIAL: NCT05997069
Title: Effects of Posterior-anterior Vertebral Mobilization Followed by Prone Press-up Exercise in Nonspecific Low Back Pain- a Randomized Controlled Trial
Brief Title: Effects of Posterior-anterior Vertebral Mobilization Followed by Prone Press-up Exercise in Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Aftab Ahmed Mirza Baig (Other)
Collaborators: Dow University of Health Sciences (Other); Sindh Institute of Physical Medicine and Rehabilitation (Other); IQRA University (Other)
Responsible Party: Sponsor-Investigator, Dr. Aftab Ahmed Mirza Baig, Principal investigator, Sindh Institute of Physical Medicine and Rehabilitation
Organization: Sindh Institute of Physical Medicine and Rehabilitation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SindhIPMR
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Low Back Pain; Chronic Low-back Pain
Keywords: lumbago; Mackenzie; movement; hot pack; thermotherapy; general stretching exercises.
MeSH Terms: conditions — Low Back Pain; Hyperthermia

STUDY DESIGN:
Intervention Model Description: In this research two groups of participants will receive different interventions.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the type of treatment. It is essential for more subjective outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Posterior-anterior vertebral mobilizations followed by Prone press-up exercise (Experimental): In experimental group the application of posterior-anterior vertebral mobilizations (three bouts of 40 seconds oscillations will be applied at the rate of approximately 3 oscillations per second and at the highest amplitude when tolerated without the reproduction of symptoms) followed by Prone press-up exercise (Ten repetitions will be performed with 5 second hold. on successful completion of 10 repetitions without increase in discomfort, second and third sets will be performed) will given.
  Interventions: Other: Posterior-anterior vertebral mobilizations followed by Prone press-up exercise
- Conventional physiotherapy (Active Comparator): In conventional physiotherapy, the application of thermotherapy on lower back region (continuous with duration of 10 minutes) by means of hot pack followed by general stretching exercises (Lower Back, Hamstring, Tensor Fasciae Latae Stretching with two sets and ten repetitions) will given.Thirty second rests will be taken every five minutes during the stretching session.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Posterior-anterior vertebral mobilizations followed by Prone press-up exercise — Posterior-anterior vertebral mobilizations of the lumbar spine are achieved by applying a force on to a spinous process in a posteroanterior direction (Back to front).
  Prone press-up exercise is started in the prone position (lying on stomach) on a flat surface. Participant keeps hands underneath the shoulders then press up his or her upper body while trying to keep the hips on the floor.
  Other Names: central vertebral mobilizations followed by prone extension exercise
  Arms: Posterior-anterior vertebral mobilizations followed by Prone press-up exercise
Other: Conventional physiotherapy — Traditionally used physiotherapy for the treatment of nonspecific low back pain (thermotherapy and general stretching exercises)
  Arms: Conventional physiotherapy

SUMMARY:
Despite advances in intervention, many patients presenting with nonspecific low back pain (NSLBP) fail to have recovery from symptoms and activity limitation. Evidence suggests that interventions commonly used by physical therapists, may be effective for some but not all subsets of people with low back pain. Posterior anterior vertebral mobilizations (PAVMs) followed by prone press up (PPU) exercise are commonly used in clinical practice without a firm evidence. Research has shown this intervention decreases nonspecific low back pain on immediate effects but there is still limitation.The objective of this study is to determine the effects of posterior anterior vertebral mobilization followed by prone press-up exercise in comparison to conventional physiotherapy in nonspecific low back pain. The hypothesis is that the PAVMs followed by PPU exercise is more effective as compared to conventional physiotherapy to improve pain, lumbar range of motion, disability and quality of life in NSLBP. So, a randomized controlled trial will be conducted at Sindh Institute of Physical Medicine and Rehabilitation. One hindered and twenty patients with 18-40 years old having NSLB will be included on the basis of non-probability and purposive sampling technique and consent will be taken. Participants will be allocated into two groups through computer random sampling software. Experimental group will receive posterior-anterior vertebral mobilization followed by prone press up exercise and control group will receive conventional therapy (thermotherapy with general stretching exercises). All participants will be assessed using assessment form. After taking demo-graphical information, pain (in standing, sitting and walking), lumbar flexion and extension, functional disability and quality of life will be assessed before and after the treatment. All the data will be analysed for descriptive and inferential analysis.

DETAILED DESCRIPTION:
Initially, sample size of 38 was calculated through open epi software version 3.01 with 95% confidence interval and 80% power of test with post-test VAS mean (4.6) and standard deviation (1.2), in experimental group 17 and post-test VAS mean (3.6) and standard deviation (0.94) in control group on the basis of previous literature. Due to the low sample size at least 50 subjects per group were considered first. After including drop rate of 20%, 60 subjects per group will be considered with sample size of 120 participants having NSLBP. A maximum drop-out rate of 20% is assumed. All the data will be kept confidential. The privacy of all patients will be maintained. The patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management will be monitored by Institutional Review Board of the same institute. Data will be analysed using SPSS 23 version. Mean ± SD will be calculated of quantitative variables like age. Frequency and percentage will be calculated for qualitative variables. Intention to treat analysis will be used. The intra-group and inter-group analysis will be performed with two way repeated measure ANOVA. The p-value of 0.025 will be considered as level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific low back pain for more than 6 weeks.
* Moderate intensity pain (3.5 -7.4 cm on Visual analogue scale)

Exclusion Criteria:

* Subject whose current symptoms of low back pain provoke, or increase, and/or peripheralize (ie, pain reported to move from the midline laterally, or to the buttocks, and/or lower extremity) with lumbar forward bending and prolonged sitting to a greater degree than with lumbar backward bending, or walking
* Any history of trauma, fracture or surgical procedure of the lumbar spine.
* Subjects administered epidural injections.
* Low back pain due to specific pathology.
* Any clinical condition that contraindicated physiotherapy intervention.
* Subjects with neurological deficits (like stroke, Parkinsonism).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity during walking on visual analogue scale | Baseline and after 15 week
  It is a self-administered 10 cm scale (line) where 0 cm suggests no pain and 10 suggests most excruciating pain. It will be used to asses pain in walking. Increase in score suggests increase in pain and decrease in score suggests decrease in pain.
Pain intensity during standing on visual analogue scale | Baseline and after 15 week
  It is a self-administered 10 cm scale (line) where 0 cm suggests no pain and 10 suggests most excruciating pain. It will be used to asses pain in standing. Increase in score suggests increase in pain and decrease in score suggests decrease in pain.
Pain intensity during sitting position on visual analogue scale | Baseline and after 15 week
  It is a self-administered 10 cm scale (line) where 0 cm suggests no pain and 10 suggests most excruciating pain. It will be used to asses pain in sitting. Increase in score suggests increase in pain and decrease in score suggests decrease in pain.
Lumbar flexion range of motion using Modified-Modified Schober test | Baseline and after 15 week
  Both posterior superior iliac spines (PSIS) of participant are marked with body marker. A midline point on sacrum (lower mark) between those two PSIS are localized and marked. Then the upper mark is marked at 15 cm above the midline point at sacrum. The distance between the marks will be measured after bending forward. The length is subtracted from 15 cm to indicate lumbar flexion range of motion. Increase in score suggests increase and decrease in score suggests decrease in flexion range of motion.
Lumbar extension range of motion using Modified-Modified Schober test | Baseline and after 15 week
  Both posterior superior iliac spines (PSIS) of participant are marked with body marker. A midline point on sacrum (lower mark) between those two PSIS are localized and marked. Then the upper mark is marked at 15 cm above the midline point at sacrum. The distance between the marks will be measured after bending backward. The change in distance between those marks indicates the lumbar extension ROM. Decrease in score suggests increase in extension and increase in score suggests decrease in extension range of motion.
Isometric endurance of back extensor muscles using prone isometric chest raise test | Baseline and after 15 week
  The test consists of assessing how many seconds the participant can keep the sternum off the floor while placed prone with the arms along the body. A small pillow is placed under the iliac crest to decrease the lumbar lordosis. The subject is asked to maintain the position for as long as possible, not exceeding a 5 min time limit.

SECONDARY OUTCOMES:
Functional disability on Oswestry Disability Index | Baseline and after 15 week
  Oswestry Disability Index questionnaire is a standard questionnaire with questions regarding pain and the disabling effect on daily activities. Its score ranges from 0 to 100 (no disability to maximum disability). decrease in score suggests decrease in disability and increase in score suggests increase in disability.
Quality of life on World Health Organization Quality of Life Brief Version | Baseline and after 15 week
  It is a self-administered questionnaire. The World Health Organization Quality of Life Brief Version (WHOQOL-BREF) addresses four quality of life domains: physical health, psychological health, social relationships and environment. The scoring is done by summing all the points of all 4 domains and transforming into 0-100 scale, where higher score means high Qquality of life and low score means low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Aftab Ahmed Mirza Baig, MSAPT, PhD, Principal Investigator — Iqra University, North Campus, Karachi; Syed Imran Ahmed, MBBS, FCPS, Study Chair — Sindh Institute of Physical Medicine and Rehabilitation
Locations (1):
- Sindh Institute Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Results will be published by the investigators in academic journals. Sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential collaborators interested in physical medicine rehabilitation and low back pain.

REFERENCES:
- [Background] Bardin LD, King P, Maher CG. Diagnostic triage for low back pain: a practical approach for primary care. Med J Aust. 2017 Apr 3;206(6):268-273. doi: 10.5694/mja16.00828. PMID 28359011
- [Background] Ganesan S, Acharya AS, Chauhan R, Acharya S. Prevalence and Risk Factors for Low Back Pain in 1,355 Young Adults: A Cross-Sectional Study. Asian Spine J. 2017 Aug;11(4):610-617. doi: 10.4184/asj.2017.11.4.610. Epub 2017 Aug 7. PMID 28874980
- [Background] Baig AAM, Ahmed SI, Ali SS, Rahmani A, Siddiqui F. Role of posterior-anterior vertebral mobilization versus thermotherapy in non specific lower back pain. Pak J Med Sci. 2018 Mar-Apr;34(2):435-439. doi: 10.12669/pjms.342.12402. PMID 29805422
- [Background] Beattie PF, Arnot CF, Donley JW, Noda H, Bailey L. The immediate reduction in low back pain intensity following lumbar joint mobilization and prone press-ups is associated with increased diffusion of water in the L5-S1 intervertebral disc. J Orthop Sports Phys Ther. 2010 May;40(5):256-64. doi: 10.2519/jospt.2010.3284. PMID 20436236
- [Background] Amjad F, Mohseni-Bandpei MA, Gilani SA, Ahmad A, Hanif A. Effects of non-surgical decompression therapy in addition to routine physical therapy on pain, range of motion, endurance, functional disability and quality of life versus routine physical therapy alone in patients with lumbar radiculopathy; a randomized controlled trial. BMC Musculoskelet Disord. 2022 Mar 16;23(1):255. doi: 10.1186/s12891-022-05196-x. PMID 35296293
- [Background] Mehyar F, Santos M, Wilson SE, Staggs VS, Sharma NK. Effect of Grade III Lumbar Mobilization on Back Muscles in Chronic Low Back Pain: A Randomized Controlled Trial. J Allied Health. 2020 Spring;49(1):20-28. PMID 32128535
- [Background] Powers CM, Beneck GJ, Kulig K, Landel RF, Fredericson M. Effects of a single session of posterior-to-anterior spinal mobilization and press-up exercise on pain response and lumbar spine extension in people with nonspecific low back pain. Phys Ther. 2008 Apr;88(4):485-93. doi: 10.2522/ptj.20070069. Epub 2008 Feb 7. PMID 18258767